CLINICAL TRIAL: NCT01667068
Title: HIV-HEART STUDY: A Prospective, Epidemiologic and Multicentre Trial to Determine the Cardiovascular Risk in HIV-infected Patients
Brief Title: Cardiovascular Diseases in HIV-infected Patients HIV-HEART Study: 7.5 Years Follow-up
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Collaborators: HIV-HEART Study Investigative Group (Unknown); German Heart Failure Network (Other); German Federal Ministry of Education and Research (Other Government); Bristol-Myers Squibb (Industry); ViiV Healthcare (Industry); Gilead Sciences (Industry); Janssen-Cilag GmbH (Unknown); Abbott (Industry); Boehringer Ingelheim (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Stefan Esser M.D., Academic Director, University Hospital, Essen
Other Study IDs: 12-4970-BO
Record Dates: First submitted 2012-08-16; First posted 2012-08-17 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Coronary Heart Disease; Heart Failure; HIV; AIDS; Metabolic Syndrome
Keywords: Cardiac Diseases; HIV-Infection; AIDS; Antiretroviral Therapy; Cardiovascular Medication; Risk Factors; coronary heart disease; heart failure; metabolic syndrome
MeSH Terms: conditions — Coronary Disease; Heart Failure; Acquired Immunodeficiency Syndrome; Metabolic Syndrome; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Regional Ruhrgebiets Cohort: HIV-positive patients in the German Ruhr-Region from out-patient clinics of hospitals and HIV-physicians pratices
  Interventions: Other: Comprehensive non invasive cardiovascular examination

INTERVENTIONS:
Other: Comprehensive non invasive cardiovascular examination — * Anamnesis with the participian
  * File recherche,Physical examination
  * Documentation of the carciovascular and antiretroviral medical therapy
  * Electrocardiogram
  * Transthoracic echocardiography
  * Exercise electrocardiogram
  * Measuring of the arterial media thickness
  * Exercise Montreal Cognitive Assesment test
  * Exercise the Grooved Pegboard test
  * Blood collection
  * Questionnaire to quality of life and health economics

SUMMARY:
Since the introduction of antiretroviral therapy life expectancy of HIV-infected persons is rising. Different cohorts are observing an increased risk for cardiovascular diseases in this aging HIV-infected population. Traditional cardiovascular risk factors like smoking are more frequent in HIV-infected persons. For example chronic inflammation due to HIV-infection and metabolic disorders also caused by some antiretroviral substances as special non-traditional risk factors in HIV-infected persons can influence the development of cardiovascular diseases additionally. Therefore new research focus in special risk profile associated with HIV-infection or antiretroviral treatment and prevention for HIV-infected patients is developing.

This present study is an ongoing prospective regional multicenter trial that was conducted to analyse the incidence, prevalence and clinical course of cardiovacular disorders in HIV-infected out-patients.

Cardiac disorders witch are associated with HIV are pericarditis, pleural effusion, pulmonary hypertension, dilated cardiomyopathy, heart failure, myocarditis, bacterial endocarditis and heart valve disorders. In addition to previously stated disorders of the heart, the premature atherosclerosis of coronary arteries, a further even more important disease of the heart in this patient population, went into the focus of most HIV-researchers and physicians.

DETAILED DESCRIPTION:
A comprehensive detailed description of the study procedures had been previously published (European Journal of medical research 2007;12:243-248).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Known HIV-infection
* Written informed consent

Exclusion Criteria:

* Acute cardiovascular disease
* Unstable hemodynamic status in the three weeks before inclusion
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participiants were included in several cities of the Ruhrarea. Locations were Essen, Bochum, Dortmund and Duisburg The study population included outpatients who were at least 18 years of age, had a known HIV-infection and exhibited a stable disease status within 4 weeks before inclusion of the trial. Written informed consent was obtained from all participants.
Sampling Method: Non-Probability Sample
Enrollment: 1481 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Diseases in HIV-infected Patients | Baseline up to 7.5 follow-up to
  The detection of prevalence, aetiology, progression and severity of cardiovascular diseases - especially of coronary artery disease in HIV-infected patients.

SECONDARY OUTCOMES:
Cardiovascular Disorders in HIV-infected Patients HIV-HEART | Baseline up to 5 years follow-up
  Complementary the study also investigates the impact of classic cardiovascular risk factors like gender, age, blood fat and also new HIV-specific risk factors of coronary artery disease like viral-load, CD4-cell count and stage of the infection. The HIV-HEART study will focus the impact of medication including cardiovascular and antiretroviral medication. Further secondary objectives will be examined, including economic costs and the subjectively quality of life of subjects with and without cardiovascular diseases in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Esser, MD, Principal Investigator — University Hospital, Essen; Till Neumann Neumann, MD, Principal Investigator — University Hospital, Essen
Locations (6):
- Germany (6):
  - University Hospital of Bochum, Department of Dermatology, Bochum
  - HIV Outpatient Department, Dortmund
  - Health Center, Duisburg
  - University Hospital, Department of Dermatology and Venerology, Essen
  - University Hospital, West German Heart Center Essen, Essen
  - Clinical Coordinating Center Leipzig, Leipzig

REFERENCES:
- [Result] Neumann T. [HIV, AIDS and the cardiovascular risk]. Internist (Berl). 2008 Apr;49(4):429-30, 432-5. doi: 10.1007/s00108-008-2049-4. German. PMID 18305915
- [Result] Reinsch N, Buhr C, Krings P, Kaelsch H, Kahlert P, Konorza T, Neumann T, Erbel R; Competence Network of Heart Failure. Effect of gender and highly active antiretroviral therapy on HIV-related pulmonary arterial hypertension: results of the HIV-HEART Study. HIV Med. 2008 Aug;9(7):550-6. doi: 10.1111/j.1468-1293.2008.00602.x. Epub 2008 Jun 28. PMID 18557952
- [Result] Reinsch N, Buhr C, Krings P, Kaelsch H, Neuhaus K, Wieneke H, Erbel R, Neumann T; German Heart Failure Network. Prevalence and risk factors of prolonged QTc interval in HIV-infected patients: results of the HIV-HEART study. HIV Clin Trials. 2009 Jul-Aug;10(4):261-8. doi: 10.1310/hct1004-261. PMID 19723613
- [Result] Neumann T, Reinsch N, Neuhaus K, Brockmeyer N, Potthoff A, Esser S, Hower M, Neumann A, Mostardt S, Gelbrich G, Erbel R; fur die HIV-HEART-Studie sowie die Kompetenznetze Herzinsuffizienz und HIV/AIDS. [BNP in HIV-infected patients]. Herz. 2009 Dec;34(8):634-40. doi: 10.1007/s00059-009-3313-7. German. PMID 20024643
- [Result] Neumann T, Esser S, Potthoff A, Pankuweit S, Neumann A, Breuckmann F, Neuhaus K, Kondratieva J, Buck T, Muller-Tasch T, Wachter R, Prettin C, Gelbrich G, Herzog W, Pieske B, Rauchhaus M, Loffler M, Maisch B, Mugge A, Wasem J, Gerken G, Brockmeyer NH, Erbel R; HIV-HEART Study Investigative Group. Prevalence and natural history of heart failure in outpatient HIV-infected subjects: rationale and design of the HIV-HEART study. Eur J Med Res. 2007 Jun 27;12(6):243-8. PMID 17666313
- [Result] Breuckmann F, Neumann T, Kondratieva J, Wieneke H, Ross B, Nassenstein K, Barkhausen J, Kreuter A, Brockmeyer N, Erbel R. Dilated cardiomyopathy in two adult human immunodeficiency positive (HIV+) patients possibly related to highly active antiretroviral therapy (HAART). Eur J Med Res. 2005 Sep 12;10(9):395-9. PMID 16183552
- [Result] Reinsch N, Kahlert P, Esser S, Sundermeyer A, Neuhaus K, Brockmeyer N, Potthoff A, Erbel R, Buck T, Neumann T. Echocardiographic findings and abnormalities in HIV-infected patients: results from a large, prospective, multicenter HIV-heart study. Am J Cardiovasc Dis. 2011;1(2):176-84. Epub 2011 Jul 30. PMID 22254197
- [Result] Lind A, Reinsch N, Neuhaus K, Esser S, Brockmeyer NH, Potthoff A, Pankuweit S, Erbel R, Maisch B, Neumann T. Pericardial effusion of HIV-infected patients ? Results of a prospective multicenter cohort study in the era of antiretroviral therapy. Eur J Med Res. 2011 Nov 10;16(11):480-3. doi: 10.1186/2047-783x-16-11-480. PMID 22027640
- [Result] Gelbrich B, Neumann T, Esser S, Potthoff A, Reinsch N, Hower M, Dannhauer KH, Loeffler M, Brockmeyer NH, Erbel R, Gelbrich G; HIV-HEART Study Investigative Group, Competence Networks Heart Failure and HIV/AIDS. Oral health and the heart - does HIV infection open a pathophysiological gateway? Int J Cardiol. 2011 Sep 1;151(2):254-7. doi: 10.1016/j.ijcard.2011.06.081. Epub 2011 Jul 18. No abstract available. PMID 21764468
- [Result] Reinsch N, Neuhaus K, Esser S, Potthoff A, Hower M, Mostardt S, Neumann A, Brockmeyer NH, Gelbrich G, Erbel R, Neumann T; German Competence Network Heart Failure; German Competence Network for HIV/AIDS. Are HIV patients undertreated? Cardiovascular risk factors in HIV: results of the HIV-HEART study. Eur J Prev Cardiol. 2012 Apr;19(2):267-74. doi: 10.1177/1741826711398431. Epub 2011 Feb 28. PMID 21450595
- [Result] Reinsch N, Neuhaus K, Esser S, Potthoff A, Hower M, Brockmeyer NH, Erbel R, Neumann T; German Competence Network for Heart Failure; German Competence Network for HIV AIDS. Prevalence of cardiac diastolic dysfunction in HIV-infected patients: results of the HIV-HEART study. HIV Clin Trials. 2010 May-Jun;11(3):156-62. doi: 10.1310/hct1103-156. PMID 20739268
- [Result] Potthoff A, Brockmeyer NH, Gelbrich G, Neuhaus K, Esser S, Reinsch N, Hower M, Mostardt S, Neumann A, Neumann T; Competence Center Cardiac Insufficiency and the Competence Network HIV/AIDS. Lipodystrophy - a sign for metabolic syndrome in patients of the HIV-HEART study. J Dtsch Dermatol Ges. 2010 Feb;8(2):92-8. doi: 10.1111/j.1610-0387.2009.07330.x. Epub 2009 Dec 14. English, German. PMID 20002869